CLINICAL TRIAL: NCT04914312
Title: Beneficial Effects of Maqui Berry Extract Combination With Omega-3 Fatty Acids on Cytokine Reduction in Elderly Obese Adults
Brief Title: Maqui Berry Extract and Omega-3 Fatty Acids for Cytokine Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00014007
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Inflammation
Keywords: maqui berry extract; omega-3 fatty acids; cytokines; blood lipids
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: randomized, controlled trial
Who Masked: Participant, Investigator
Masking Description: Experimental capsules matched to placebo capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maqui berry extract and omega-3 fatty acids (Experimental): 2 capsules BID per day containing a total of 600 mg of Maqui extract; 4 capsules per day supplying a total of 2000 mg EPA and 1000 mg DHA
  Interventions: Dietary Supplement: Maqui berry/omeg-3 fatty acids
- Control (Placebo Comparator): 4 olive oil soft gelatin capsules and inert two-piece capsules containing maltodextrin
  Interventions: Dietary Supplement: Placebos

INTERVENTIONS:
Dietary Supplement: Maqui berry/omeg-3 fatty acids — 2 capsules BID per day containing a total of 600 mg of Maqui extract; 4 capsules per day supplying a total of 2000 mg EPA and 1000 mg DHA
  Arms: Maqui berry extract and omega-3 fatty acids
Dietary Supplement: Placebos — 4 olive oil soft gelatin capsules and inert two-piece capsules containing maltodextrin
  Arms: Control

SUMMARY:
The purpose of this trial is to determine the effect of maqui extract plus omega-3 fatty acids compared to a placebo for reducing inflammatory cytokine levels in older, obese adults.

DETAILED DESCRIPTION:
Anthocyanins, a subclass of flavonoids, are plant pigments that provide the rich color of many plants, fruits, and flowers. Health benefits of anthocyanins have been widely reported in the research literature, particularly for disease conditions associated with oxidative stress, such as cardiovascular and neurodegenerative diseases. Emerging evidence suggests that anthocyanins may also modulate gut microbiota, which can impact a wide variety of health conditions. Maqui berries (Aristotelia chilensis), indigenous to Chile, have one of the highest concentrations of anthocyanins in the plant world; moreover, the dominant anthocyanin in maqui berries is delphinidin. Delphinidin is more bioavailable than most flavonoids, with intact molecules absorbed in appreciable amounts in less than an hour after consumption. Systemic effects of delphinidin include reduced inflammation due to downregulation of NF-kB, the transcription factor that initiates the generation of pro-inflammatory cytokines. The omega-3 fatty acid eicosapentaenoic acid [EPA], a component of omega-3 fatty acid concentrates, also has anti-inflammatory properties. There is much empirical evidence demonstrating beneficial effects of EPA supplementation, linked mainly to reductions in inflammation. It has been demonstrated the dietary supplementation with EPA-rich marine oil concentrations reduces cytokine levels up to 15%.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 50-85 years old
* Generally healthy, non-smoker
* Able to provide informed consent
* BMI: 30-40 kg/m2

Exclusion Criteria:

* Existing auto-immune conditions
* Use of warfarin or other blood thinners
* Use of anti-inflammatory drugs, cardiovascular medications, lipid-altering drugs, and hormone replacement therapy
* Individuals engaged in vigorous exercise (>2 x 30 min/week), vegetarians, and people who routinely take multivitamins or herbal supplements.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | change from baseline at day 56
  Blood concentrations of IL-6
Interleukin-1 beta (IL-1 beta) | change from baseline at day 56
  Blood concentration of IL-1 beta
Tumor Necrosis Factor (TNF) | change from baseline at day 56
  Blood concentration of TNF

SECONDARY OUTCOMES:
Arachidonic acid (AA) | change from baseline at day 56
  Blood concentration of AA
Eicosapentaenoic acid (EPA) | change from baseline at day 56
  Blood concentration of EPA

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No